CLINICAL TRIAL: NCT00313885
Title: Efficacy and Safety of SR46349B (1 and 5mg/Day) Administered During 8 Weeks in Patients With Sleep Disorders in Fibromyalgia: Multi-center, Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Efficacy and Safety of SR46349B in Patients With Sleep Disorders in Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT5400
Record Dates: First submitted 2006-04-07; First posted 2006-04-12 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Fibromyalgia; Sleep; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — SR 46349B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): 1 mg daily
  Interventions: Drug: eplivanserin (SR46349)
- 2 (Experimental): 5 mg daily
  Interventions: Drug: eplivanserin (SR46349)
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: eplivanserin (SR46349) — oral administration
  Arms: 1; 2
Drug: placebo — oral administration
  Arms: 3

SUMMARY:
Fibromyalgics frequently report sleep disturbances, in particular poor and unrefreshing sleep. Additionally, studies have reported that sleep problems, pain and mood disturbances are associated in patients with fibromyalgia. By improving the quality of sleep, complaints of poor and unrefreshing sleep, fatigue, pain, which are among the main components of this chronic pain disorder may be improved.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate the effectiveness and safety of 2 doses of the investigational product in subjects with sleep disorders with fibromyalgia as compared to placebo (a substance which contains no active ingredient). The study will last approximately 70 days and will include 7 office visits.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must fulfill the diagnosis criteria of fibromyalgia according to the American College of Rheumatology
* Based on patient's information:
* The patient must complain of unrefreshing sleep for at least 3 nights per week over the past month.
* The patient spends at least 6.5 hours and not more than 9 hours, in bed, each night over the past 2 weeks.
* Female patients of childbearing potential must have a confirmed negative pregnancy test at the end of the screening period and use an acceptable method of birth control throughout the study
* Written, signed and dated informed consent must be obtained from each patient
* Willing to abstain from taking any medication or treatment prohibited as per the protocol

Exclusion Criteria:

* Females who are lactating or pregnant
* Night shift workers, and individuals who nap 3 or more times per week over the preceding month (nap: intentionally sleeping for more than 20 minutes during the day).
* Consumption of beverage with caffeine (i.e. tea, coffee, or cola) comprising more than 2 cups or glasses per day
* Past or Current medical history of any significant, severe, or unstable acute or chronically progressive medical or surgical disorder which may affect patient safety

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
refreshing quality of sleep measured by the patient sleep questionnaire | 8 weeks

SECONDARY OUTCOMES:
sleep parameters (maintenance, duration, induction and quality) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (12):
- United States (11):
  - Radiant Research, Phoenix, Arizona
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Miami Research Assoc., Inc., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Comprehensive Neuroscience, Atlanta, Georgia
  - Physicians Research Group, Indianapolis, Indiana
  - Wichita Clinic PA, Wichita, Kansas
  - Westroads Medical Group, Omaha, Nebraska
  - Physicians Research Options, Ogden, Utah
  - Seattle Rheumatology Assoc., Seattle, Washington
- Sanofi-Aventis Administrative Office, Laval, Canada